CLINICAL TRIAL: NCT00778544
Title: Randomized, Open-Label, 2 - Way Crossover, Bioequivalence Study of Amoxicillin-Clavulanic Acid 600 mg- 42.9 mg/ 5 mL Oral Suspension and Augmentin ES-600 (Reference) Following a 600 mg- 42.9 mg Dose in Healthy Subjects Under Fed Conditions.
Brief Title: Bioequivalence Study of Amoxicillin-Clavulanic Acid 600 mg-42.9 mg/ 5 mL Oral Suspension Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 60250
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence amoxicillin-clavulanic acid 600 mg 42.9 mg per 5 mL oral suspension
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): amoxicillin-clavulanic acid 600 mg- 42.9 mg/ 5 mL oral suspension of Ranbaxy
  Interventions: Drug: amoxicillin-clavulanic acid 600 mg- 42.9 mg/ 5 mL oral suspension
- 2 (Active Comparator): Augmentin ES-600
  Interventions: Drug: amoxicillin-clavulanic acid 600 mg- 42.9 mg/ 5 mL oral suspension

INTERVENTIONS:
Drug: amoxicillin-clavulanic acid 600 mg- 42.9 mg/ 5 mL oral suspension

SUMMARY:
The objective of this study was to compare the rate and extent of absorption of Ranbaxy Laboratories Limited, India, Amoxicillin-Clavulanic acid and GlaxoSmithKline, U.S.A. (Augmentin ES-600), amoxicillin-clavulanic acid, administered as a 1 x 5 mL (600 mg - 42.9 mg) oral suspension, under fed conditions.

DETAILED DESCRIPTION:
This was a single center, randomized, single-dose, open label, 2 - way crossover bioequivalence study to compare the rate and extent of absorption of a test amoxicillin-clavulanic acid versus Augmentin ES-600, a reference amoxicillin- clavulanic acid, under fed conditions. Prior to the study commencement, subjects were randomly assigned to a treatment in accordance with the randomization scheme generated by Anapharm. Subjects were confined to the Anapharm Clinical research Facility from at least 11 hours prior to drug administration until after the 12.0 hour post-dose blood draw, in each period. The treatment phases were separated by a washout period of 14 days.

A total of sixty-two (62) healthy adult subjects signed the study specific informed consent form and were confined for period I; of these subjects forty eight (48), (21 males and 27 females) were enrolled and dosed in the study; forty six (46) of these enrolled subjects completed the clinical phase of the study

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in this study will be members of the community at large. The recruitment advertisements may use various media types (e.g. radio, newspaper, SFBP Anapharm Web site, SFBC Anapharm Volunteers database). Subjects must meet all of the following criteria to be included in the study:

  1. Male or female, smoker or non-smoker, 18 years of age or older
  2. Capable of consent
  3. BMI greater than or equal to 19.0 and less than 30.0

Exclusion Criteria:

* Subjects to whom any of the following applies will be excluded from the study:

  1. Clinically significant illness or surgery within 4 weeks prior to dosing
  2. Any clinically significant abnormality or abnormal laboratory test results found during medical screening
  3. Any reason which in the opinion of the clinical Sub-Investigator, would prevent the subject from participating in the study
  4. Positive tests for hepatitis B, hepatitis C, or HIV at screening
  5. ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mm Hg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening
  6. History of significant alcohol abuse or drug abuse within one year prior to the screening visit
  7. Regular use of alcohol within six months prior to the screening visit (more than 14 units of alcohol per week [ 1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol])
  8. Use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to screening
  9. History of allergic reactions to amoxicillin-clavulanic acid, penicillin, or other related drugs
  10. Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, Omeprazole; examples of inhibitors: antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolines, antihistamines) within 30 days prior to administration of the study medication
  11. Use of an investigational drug or participation in an investigational study within 30 days prior to dosing
  12. Clinically significant history or presence of any gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
  13. Any clinically significant history or presence of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, or metabolic disease.
  14. Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to the administration of the study medication, except for topical products without systemic absorption and hormonal contraceptives
  15. Difficulty to swallow study medication
  16. Smoking more than 25 cigarettes per day
  17. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Clinical Sub-Investigator, could contraindicate the subject's participation in this study
  18. A depot injection or an implant of any drugs (other than hormonal contraceptives) within 3 months prior to administration of study medication
  19. Donation of plasma (500 mL) within 7 days prior to the drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:

      * 50 mL to 499 mL of whole blood within 30 days
      * More than 499 mL of whole blood within 56 days prior to the drug administration
  20. Wear of dentures or presences of braces at the time of dosing or any piercing in mouth, lips, and/ or tongue
  21. Positive urine pregnancy test at screening
  22. Breast feeding subject
  23. Female subjects of childbearing potential having unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration. Hormonal contraceptives are permitted during the study but are not an acceptable method of contraception. Acceptable methods of contraceptives are:

      * Intra-uterine contraceptive device (placed at least 4 weeks prior to study drug administration
      * Condom or diaphragm + spermicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-06; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Anapharm, Québec, Quebec, Canada

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html